CLINICAL TRIAL: NCT02182141
Title: An Open Label Dose Escalation Study of BIBF 1120 Administered Orally for Four Weeks in Patients With Relapsed or Refractory Multiple Myeloma With Repeated Administration in Patients With Clinical Benefit
Brief Title: An Dose Escalation Study of BIBF 1120 Administered in Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1199.2
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

ARMS (1):
- BIBF 1120 (Experimental)
  Interventions: Drug: BIBF 1120 ES

INTERVENTIONS:
Drug: BIBF 1120 ES

SUMMARY:
Maximum tolerated dose (MTD), safety, pharmacokinetics, efficacy of BIBF 1120, pharmacodynamics

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed diagnosis of multiple myeloma, who did not respond to or relapsed after either anthracyclines and pulsed glucocorticoids or high-dose therapy and who are currently not eligible for transplant modalities.
2. Age 18 years or older
3. Life expectancy of at least six months
4. Patients have to give written informed consent (which must be consistent with ICH-GCP and local legislation)
5. Eastern Cooperative Oncology Group (ECOG) performance score <2.
6. Recovery from all therapy-related toxicities from previous chemo-, immuno- or radiotherapies.

Exclusion Criteria:

1. History of relevant surgical procedures during the last four weeks prior to treatment with the trial drug, or active ulcers, fractures or injuries with incomplete healing
2. Active infectious disease
3. Uncontrolled, severe hypertension
4. Gastrointestinal disorders anticipated to interfere with the resorption of the study drug
5. Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the protocol
6. Absolute neutrophil count less than 1000 / mm³.
7. Platelet count less than 30 000 / mm³
8. Conjugated Bilirubin greater than 2 mg / dl (> 34 μmol/L, SI unit equivalent)
9. Aspartate amino transferase (AST) and / or alanine amino transferase (ALT) greater than three times the upper limit of normal
10. Endogenous creatinine clearance (ECC) <20 ml/min
11. Women and men who are sexually active and unwilling to use a medically acceptable method of contraception
12. Pregnancy or breastfeeding
13. Treatment with other investigational drugs or participation in another clinical trial within the past four weeks before start of therapy or concomitantly with this trial (except for present trial drug)
14. Patients unable to comply with the protocol
15. Active alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2003-04; Primary Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 11 months

SECONDARY OUTCOMES:
Incidence and intensity of adverse events according to Common Toxicity Criteria (CTC) associated with increasing doses of BIBF 1120 | Up to 11 months
Change from baseline in laboratory parameters | Baseline, up to 11 months
Objective tumor response in surrogate markers | Baseline, up to 11 month
Concentration at 2h (C2,1) | 2 hours after first administration
Change from baseline in cellular protein tyrosine kinase inhibition | Baseline, up to 11 months
Change from baseline in Eastern Cooperative Oncology Group (ECOG) performance score | Baseline, up to 11 months
Change in vital signs | up to 11 months
Change from baseline in electrocardiogram (ECG) | Baseline, up to 11 months
Predose concentration immediately before administration of the Nth dose over the dosing interval τ (Cpre,N) | Up to day 28
Area under the plasma concentration-time curve during the dosing interval τ (24 h) at steady state (AUCτ,ss) | Up to 11 months
Plasma concentration at the time point immediately before dosing at steady state (Cpre,ss) | Up to 11 months
Minimum plasma concentration during the dosing interval τ at steady state (Cmin,ss) | Up to 11 months
Maximum plasma concentration during the dosing interval τ at steady state (Cmax,ss) | Up to 11 months
Time to reach minimum plasma concentration during the dosing interval τ at steady state (tmin,ss) | Up to 11 months
Time to reach maximum plasma concentration during the dosing interval τ at steady state (tmax,ss) | Up to 11 months
Terminal half-life at steady state (t1/2,ss) | Up to 11 months
Apparent plasma clearance at steady state (CL/F,ss) | Up to 11 months
Mean residence time at steady state (MRTpo,ss) | Up to 11 months
Apparent volume of distribution during the terminal phase at steady state (Vz/F,ss) | Up to 11 months
Tumor response assessed according to the European Group for Blood and Marrow Transplantation (EBMT) criteria | Up to 11 months